CLINICAL TRIAL: NCT06065137
Title: Standardised Drug Provocation Testing in Perioperative Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-5451; 3265 (Other: EDGE)
Record Dates: First submitted 2023-09-19; First posted 2023-10-03 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Allergic Reaction; Hypersensitivity; Perioperative Complication; Anaphylaxis; Anaphylactic Reaction; Immediate Hypersensitivity; Hypersensitivity, Drug
MeSH Terms: conditions — Hypersensitivity; Anaphylaxis; Hypersensitivity, Immediate; Drug Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- POH patients (Experimental): incremental administration of investigated anesthetics up to full therapeutic dose in POH patients.
  Interventions: Diagnostic Test: Full dose DPT with propofol; Diagnostic Test: Full dose DPT with ketamine; Diagnostic Test: Full dose DPT with etomidate; Diagnostic Test: Full dose DPT with midazolam; Diagnostic Test: Full dose DPT with fentanyl; Diagnostic Test: Full dose DPT with sufentanyl; Diagnostic Test: Full dose DPT with alfentanil; Diagnostic Test: Full dose DPT with remifentanil; Diagnostic Test: Full dose DPT with rocuronium; Diagnostic Test: Full dose DPT with atracurium; Diagnostic Test: Full dose DPT with cisatracurium; Diagnostic Test: Full dose DPT with succinylcholine

INTERVENTIONS:
Diagnostic Test: Full dose DPT with propofol — Incremental administration of propofol up to a cummulative full therapeutic dose (2mg/kg) in POH patients investigated for propofol. Doses will be administered every 15 minutes starting at 1/100th of the dose, followed by 1/10th of the dose, 3/10th of the dose and ultimately 6/10th of the dose (0.02mg/kg-0.2 mg/kg -0.6 mg/kg -1.2mg/kg).
Diagnostic Test: Full dose DPT with ketamine — Incremental administration of ketamine up to a cummulative full therapeutic dose (1mg/kg) in POH patients investigated for ketamine. Doses will be administered every 15 minutes starting at 1/100th of the dose, followed by 1/10th of the dose, 3/10th of the dose and ultimately 6/10th of the dose (0.01 mg/kg -0.1 mg/kg -0.3 mg/kg -0.6mg/kg).
Diagnostic Test: Full dose DPT with etomidate — Incremental administration of etomidate up to a cummulative full therapeutic dose (0.2mg/kg) in POH patients investigated for etomidate. Doses will be administered every 15 minutes starting at 1/100th of the dose, followed by 1/10th of the dose, 3/10th of the dose and ultimately 6/10th of the dose (0.002 mg/kg -0.02 mg/kg -0.06 mg/kg -1.2mg/kg).
Diagnostic Test: Full dose DPT with midazolam — Incremental administration of midazolam up to a cummulative full therapeutic dose (0.05mg/kg) in POH patients investigated for midazolam. Doses will be administered every 15 minutes starting at 1/100th of the dose, followed by 1/10th of the dose, 3/10th of the dose and ultimately 6/10th of the dose (0.0005 mg/kg -0.005 mg/kg -0.015 mg/kg -0.03mg/kg).
Diagnostic Test: Full dose DPT with fentanyl — Incremental administration of fentanyl up to a cummulative full therapeutic dose (1mcg/kg) in POH patients investigated for fentanyl. Doses will be administered every 15 minutes starting at 1/100th of the dose, followed by 1/10th of the dose, 3/10th of the dose and ultimately 6/10th of the dose (0.01 mcg/kg -0.1 mcg/kg -0.3 mcg/kg -0.6mcg/kg).
Diagnostic Test: Full dose DPT with sufentanyl — Incremental administration of sufentanyl up to a cummulative full therapeutic dose (0.1mcg/kg) in POH patients investigated for sufentanyl. Doses will be administered every 15 minutes starting at 1/100th of the dose, followed by 1/10th of the dose, 3/10th of the dose and ultimately 6/10th of the dose (0.001 mcg/kg -0.01 mcg/kg -0.03 mcg/kg -0.06µg/kg).
Diagnostic Test: Full dose DPT with alfentanil — Incremental administration of alfentanil up to a cummulative full therapeutic dose (10mcg/kg) in POH patients investigated for alfentanil. Doses will be administered every 15 minutes starting at 1/100th of the dose, followed by 1/10th of the dose, 3/10th of the dose and ultimately 6/10th of the dose (0.1 mcg/kg -1 mcg/kg -3 mcg/kg -6µg/kg).
Diagnostic Test: Full dose DPT with remifentanil — Incremental administration of remifentanil up to a cummulative full therapeutic dose (0.5mcg/kg) in POH patients investigated for remifentanil. Doses will be administered every 15 minutes starting at 1/100th of the dose, followed by 1/10th of the dose, 3/10th of the dose and ultimately 6/10th of the dose (0.005 mcg/kg -0.05 mcg/kg -0.15 mcg/kg -0.3µg/kg).
Diagnostic Test: Full dose DPT with rocuronium — Incremental administration of rocuronium up to a cummulative full therapeutic dose (0.6mg/kg) in POH patients investigated for rocuronium. Doses will be administered every 15 minutes starting at 1/100th of the dose, followed by 1/10th of the dose (0.006 mg/kg -0.06 mg/kg ). In a second session 3/10th of the dose and ultimately 7/10th of the dose (0.18 mg/kg -0.42mg/kg) are administerd under general anesthesia.
Diagnostic Test: Full dose DPT with atracurium — Incremental administration of atracurium up to a cummulative full therapeutic dose (0.5mg/kg) in POH patients investigated for atracurium. Doses will be administered every 15 minutes starting at 1/100th of the dose, followed by 1/10th of the dose (0.005 mg/kg -0.05 mg/kg ). In a second session 3/10th of the dose and ultimately 7/10th of the dose (0.15 mg/kg -0.35mg/kg) are administered under general anesthesia .
Diagnostic Test: Full dose DPT with cisatracurium — Incremental administration of cisatracurium up to a cummulative full therapeutic dose (0.15mg/kg) in POH patients investigated for cisatracurium. Doses will be administered every 15 minutes starting at 1/100th of the dose, followed by 1/10th of the dose (0.0015 mg/kg -0.015 mg/kg ). In a second session 3/10th of the dose and ultimately 7/10th of the dose (0.045 mg/kg -0.105mg/kg) are administered under general anesthesia .
Diagnostic Test: Full dose DPT with succinylcholine — Incremental administration of succinylcholine up to a cummulative full therapeutic dose (1mg/kg) in POH patients investigated for succinylcholine. Doses will be administered every 15 minutes starting at 1/100th of the dose, followed by 1/10th of the dose (0.01 mg/kg -0.1 mg/kg). In a second session 3/10th of the dose and ultimately 7/10th of the dose (0.3 mg/kg -0.7mg/kg) are administered under general anesthesia.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and outcome of systematic drug provocation testing with anaesthetics at therapeutic doses in adult patients undergoing diagnostic work-up for perioperative hypersensitivity.

DETAILED DESCRIPTION:
Perioperative hypersensitivity reactions (POH) pose a risk for major morbidity and mortality in the perioperative period. After resolution of the initial reaction it is crucial to determine the culprit drug to allow safe anaesthetics for future procedures.However this is not easy, as many drugs are administered near simultaneously and both anaesthesia and surgery may provoke or mask many of the symptoms of a hypersensitivity reaction. Conventional testing seems to offer good predictive value based on the low incidence of POH in subsequent re-exposures after negative work-up. Despite negative work-up anaesthetists often chose not to re-administer an neuromuscular blocking agent (NMBA) used in the index reaction, especially if no other culprit was found. This introduces an important bias as this group (no culprit found, NMBA not re-exposed) might be at the highest risk of containing false negatives as NMBA are the most frequent cause of POH in our region.The same remark can be made regarding earlier attempts by our group and others at establishing the negative predictive value (NPV) of conventional testing through retrospective analysis of subsequent re-exposures.To truly establish the NPV for conventional testing and thus the need for DPT, a prospective approach is needed where all patients are challenged with index drugs after negative conventional testing.

Adult patients that are referred for diagnostic work-up for POH will be included if they have a clinical history fitting with POH.

All patients will first receive a full diagnostic work-up for all index products consisting of in vivo (skin tests) and in vitro (specific IgE and -for drugs in which it is available- basophil activation tests). Clinical reactions (both index reactions and any reactions during DPT) will be classified according to the National Audit Program (NAP-6) classification which separates non-fatal POH in 4 grades:

* NAP 1 (only cutaneous/mucosal signs)
* NAP 2 (circulatory or respiratory symptoms which don't require treatment)
* NAP 3 (circulatory or respiratory symptoms which require treatment or potential airway compromise)
* NAP 4 (fulfilling indications for cardiopulmonary resuscitation)

Skin tests will be performed at the allergology day clinic following the protocols of the French Society for Anaesthesia and Intensive Care and the French Society of Allergology. Based on these results we make a distinction between patients with an identified culprit and those without an identified culprit.

If a culprit has been found, all other index drugs are challenged at therapeutic doses. The standard testing is performed for alternatives for the culprit drug in the same drug class (such as NMBA) and one drug from this class that tests negative is also used in a challenge at a therapeutic dose.

If no culprit has been found after the initial work-up of skin tests and in vitro tests the next step is determined by the severity of the initial reaction. In NAP-6 grade 1-3 reactions all index drugs are challenged at therapeutic doses. As the benefits of DPT have yet to be fully quantified the risk-benefit analysis in the most severe reactions (NAP 4) is difficult to make. Hence, we use an 'confirmation by elimination' principle in these cases in which we only challenge with the drugs that do not carry the highest likelihood of being the culprit. This likelihood is based on both timing and epidemiology as NMBA are a much more common cause of POH in our region than all other anaesthetics combined. By eliminating all other drugs we 'clear' them for future use and gain confidence in our suspicion of the most likely culprit without having to administer them in this population.

ELIGIBILITY:
Inclusion Criteria:

* patients consulting the allergology department of the Antwerp University hospital medical with a history consistent with perioperative hypersensitivity
* Indication for diagnostic work-up as determined at an interdisciplinary meeting between allergologists and anaesthetists
* willing to sign separate informed consent forms for both general anaesthesia and the Drug Provocation Test.

Exclusion Criteria:

* patient refusal
* incomplete diagnostic work-up
* history inconsistent with perioperative hypersensitivity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Hypersensitivity during DPT | 1 hour
  Prevalence of hypersensitivity during direct provocation for drugs that tested negatively in conventional tests.

SECONDARY OUTCOMES:
Severe reactions during DPT | 1 hour
  Prevalence of severe (NAP 3-4) hypersensitivity reactions during direct provocation testing
Adverse events during DPT | 1 hour
  Prevalence of adverse events during or after direct provocation testing
Sensitivity of conventional tests | 1 hour
  Sensitivity of skin tests, specific IgE and basophil activation tests for anaesthetics

CONTACTS AND LOCATIONS:
Overall Officials: Vera Saldien, MD,PhD, Principal Investigator — University Hospital Antwerp, Head of department of anesthesiology
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium